CLINICAL TRIAL: NCT04664218
Title: Are You in a Poor Country; HIPEC is Still in Reach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed I Abdelhamid, Associate professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HIPEC is still in reach 2020
Record Dates: First submitted 2020-10-24; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: HIPEC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with Peritoneal carcinomatosis (Experimental): Peritoneal carcinomatosis (PC) is a well-known sequel of multiple abdominal malignancies either arising from the gastro-intestinal tract or of gynaecologic origin. On occurrence, PC is mostly considered as a very bad prognostic sign hence it affects the overall survival with very poor response to systemic chemotherapy.
  Interventions: Device: HIPEC device

INTERVENTIONS:
Device: HIPEC device — To report the affordability on using the HIPEC machine of our design compared to the standard ones in poor places.

SUMMARY:
Peritoneal carcinomatosis (PC) is a well-known sequel of multiple abdominal malignancies either arising from the gastro-intestinal tract or of gynaecologic origin. On occurrence, PC is mostly considered as a very bad prognostic sign hence it affects the overall survival with very poor response to systemic chemotherapy.

On introduction of the new concept of combined optimal cytoreduction (CRS) followed by hyperthermic intraperitoneal chemotherapy (HIPEC), promising prognosis began to be shown.

A major obstacle which may face application of HIPEC manoeuvre is the cost either of the machine or the disposable kit used in handling the chemotherapy, heating it and delivering it to the patient, hence we established our machine design with its disposable kits making it available for use in poor places.

DETAILED DESCRIPTION:
As aforementioned the use of HIPEC technique offered a promising results in dealing with peritoneal carcinomatosis the high costs seems to be a considerable obstacle in some poor places so we inented a machine with considerably lower costs both in the machine composition and its disposable kit used for every patient we used it for six years in a trial to find any shortage, obstacles or any technical, therapeutic or financial drawbacks compared to the published data of the standard machines

ELIGIBILITY:
Inclusion Criteria:

* Any patient candidate for HIPEC procedure

Exclusion Criteria:

* Contraindications to HIPEC procedure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Thermal efficiency of the machine | 6 years of the study using the machine
  The ability of the machine to warm the chemoperfusate to 43 c for 90 minutes (the duration of peritoneal perfusion)
Electrical efficiency of the machine | 6 years of the study using the machine
  Reporting any interruption or unexplained stop of the thermostat resulting in stopping of chemoperfusate flow to and out of the abdomen during the 90 minutes of the maneuver
The manufacturing costs in US dollar | one weak at the start of the trial
  the costs paid by the owner of manufacturing the machine throughout collecting its components and technical fitting them into a machine
The disposable costs in US dollar | 6 years of the study using the machine
  the costs spent by the patient at each use paid for the disposable parts of the machine of the chemotherapy perfusion circuit to and from the patient

SECONDARY OUTCOMES:
Adverse effects on the patient following HIPEC | 4 weeks
  following the patient in the postoperative period searching for adverse effects of HIPEC resulting from either the chemotherapy used or the physical activity of the machine